CLINICAL TRIAL: NCT00267865
Title: AIDS-Related Primary Central Nervous System Lymphoma: A Phase II Pilot Study of High-Dose Intravenous Methotrexate With Rituximab Leucovorin Rescue and Highly Active Antiretroviral Therapy
Brief Title: Chemotherapy and HAART to Treat AIDS-related Primary Brain Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060051; 06-C-0051; NCT00304044 (obsolete NCT alias)
Record Dates: First submitted 2005-12-21; First posted 2005-12-21 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: AIDS-Related-Primary Central Nervous System Lymphoma
Keywords: Human immunodeficiency virus; Acquired immunodeficiency syndrome; High Dose Methotrexate; Methotrexate; Rituximab; CNS Lymphoma; Central Nervous System Lymphoma; AR-PCNSL; Epstein-Barr virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Epstein-Barr Virus Infections | interventions — Methotrexate; Rituximab; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab, High-Dose Methotrexate & Leucovorin Treatment (Experimental): Induction treatment cycles with rituximab, high-dose methotrexate and leucovorin will be administered every 2 weeks for 6 cycles. Two additional consolidation cycles of high-dose methotrexate without rituximab will be administered at 4 weeks and 8 weeks following completion of the combined therapy.
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Leucovorin

INTERVENTIONS:
Drug: Methotrexate — 6000 mg/m^2 will be administered by intravenous infusion over 4 hours after confirming that the recipient patients urine pH is within the range greater than or equal to 7 to less than or equal to 8, and urine output is greater than or equal to 100 mL/hour.
  Other Names: Xatmep; Trexall; Otrexup (PF); Rasuvo
Drug: Rituximab — 375 mg/m^2 intravenous (IV) day 1 of each cycle prior to administration of high-dose methotrexate
  Other Names: Rituxan; MabThera
Drug: Leucovorin — Leucovorin calcium doses will be administered orally or by short intravenous (IV) infusion over 15 minutes
  Other Names: Folinic acid; citrovorum factor

SUMMARY:
This study will investigate the use of chemotherapy plus highly active antiretroviral therapy (HAART) in patients with Acquired Immunodeficiency Syndrome (AIDS)-related primary brain lymphoma. None of the drugs used in this study are experimental, but chemotherapy plus HAART has not been established as a standard treatment in patients with AIDS. The chemotherapy regimen used in this study (see below) was chosen because it may be less toxic to immune cells called T-lymphocytes than most drug treatments for lymphoma.

People with AIDS 18 and older and have primary brain lymphoma may be eligible for this study. Candidates are screened with a medical history and physical examination, magnetic resonance imaging (MRI), computed tomography (CT) and positron emission tomography (PET) scans, cerebrospinal fluid studies, brain biopsy at tumor sites, if possible, electrocardiogram and blood tests.

Participants undergo six 2-week "induction treatment" cycles of HAART plus chemotherapy with methotrexate, rituximab and leucovorin, followed by two 4-week "consolidation" treatment cycles using HAART, methotrexate and leucovorin, and then HAART alone. Rituximab is given by intravenous (intravenous (IV), through a vein) day 1 of each cycle. Also on day 1 IV fluids are given to lower acidity in the urine to protect the kidneys from the methotrexate. On day 2, methotrexate is infused through a vein over 4 hours. Starting 24 hours after initiation of the methotrexate infusion, leucovorin is given every 3 to 6 hours (first IV and then possibly by mouth) until the drug decreases to a target level in the blood. HAART is begun as soon as possible. The specific HAART regimen for each patient is determined individually. All patients are hospitalized the first week of every 2-week treatment cycle for safety monitoring. In addition to HAART and chemotherapy, patients undergo the following tests and procedures:

* Intellectual functioning: Before starting treatment, patients are tested for their ability to understand basic concepts and coordination in order to be able to evaluate how the brain lymphoma affects thinking and concentration. After the lymphoma appears to have resolved, more formal and intensive tests are done. The intensive tests are repeated each year, and shorter, interim tests are done about every 6 months. Also, a specialist periodically monitors patients' understanding of HAART and the importance of this therapy.
* Blood tests: Blood is drawn every day during hospitalizations to measure methotrexate levels and to evaluate kidney and liver function and blood counts. Blood is also drawn before starting therapy, when the lymphoma disappears, 6 months after completing treatment, and any time it appears that the lymphoma may have recurred to test for Epstein-Barr virus (EBV), a virus that is almost always present in AIDS-related primary brain lymphoma.
* Imaging tests: Patients undergo magnetic resonance imaging (MRI) and positron emission tomography (PET) scans periodically to monitor the effects of treatment on the lymphoma. MRI scans are done after the 2nd, 4th, 6th, and 8th treatments, then every 2 months for three times, every 3 months for six times, every 6 months for four times, and then every year for 5 years, or sooner if there is a concern about the brain. PET scans are done after the first cycle, after the MRI suggests the lymphoma is gone, and then yearly.
* Lumbar puncture (spinal tap): This test is done to look for EBV in the cerebrospinal fluid (CSF). Under local anesthetic, a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord and a small amount of fluid is collected through the needle. This test is done at the same times as the blood tests for EBV.
* Eye examinations: Patients' eyes are examined periodically because brain lymphoma can sometimes spread to the eye and because some people with AIDS-related primary brain lymphoma are at risk of certain eye infections.

DETAILED DESCRIPTION:
Background: Acquired Immunodeficiency Syndrome (AIDS)-related primary central nervous system lymphoma (AR-PCNSL) is an Epstein-Barr virus (EBV)-driven lymphoproliferative process that typically results in death within a few months. Essentially all of the cases are immunoblastic cluster of differentiation 20 (CD20+) tumors, and occur once the cluster of differentiation 4 (CD4+) cells have fallen to below 50 cells/mm^3. Highly active antiretroviral therapy (HAART) can result in immune reconstitution that decreases the risk of AR-PCNSL. However, a subset of human immunodeficiency virus (HIV)-infected patients still develops ARPCNSL, often because they are unaware that they are HIV infected, or they do not take HAART. Treatment options for such patients are limited. In the non-AIDS setting, chemotherapy has become the standard of care for primary central nervous system lymphoma (PCNSL) and late neurocognitive decline consequent to radiotherapy can be avoided by such approaches. In the pre-HAART era, AR-PCNSL was generally treated with whole brain radiotherapy, however death due to recurrent lymphoma or to other AIDS complications occurred prior to the potential manifestations of late occurring radiation-related neurotoxicity. Radiation-sparing approaches have not been studied in AR-PCNSL in the HAART era, where advances in antiretroviral therapy have made curative intent chemotherapy feasible for most patients with HIV infection.

Objectives: The primary objective of this study is to estimate the fraction of patients with AR-PCNSL receiving experimental treatment consisting of HAART, combined with rituximab, high-dose methotrexate and leucovorin (R-HD-MTX) who are alive and without recurrent lymphoma or severe cognitive problems at two years. .

Eligibility: HIV-infected, age 18 years or older, AR-PCSNL that has not previously been treated, and be able to give informed consent or have a durable power of attorney who can provide informed consent, HIV profile that makes them likely to respond to HAART. There are a number of other specific inclusion and exclusion criteria, in part to exclude patients who would be unlikely to tolerate the therapy.

Design: Phase II pilot study investigating R-HD-MTX given with leucovorin rescue and HAART as a treatment for AR-PCNSL. Evaluation will include quantitative measurement of lymphocyte subsets, quantitative polymerase chain reaction (PCR) of HIV and EBV viral loads (including both blood and cerebrospinal fluid in the case of EBV) to assess immune response and anti-viral effects. Tumor evaluation with brain magnetic resonance imaging (MRI) and brain fluoro-2-deoxy-d-glucose positron emission tomography (FDG-PET scans) will be used for staging and response assessment. Longitudinal neuropsychologic testing after complete responses are documented will serve to evaluate neurocognitive parameters post therapy.

a separate cohort for additional secondary endpoints.

ELIGIBILITY:
* INCLUSION CRITERIA:

Positive human immunodeficiency virus (HIV) serology (previous records acceptable)

* Diagnosis of Primary Central Nervous System Lymphoma
* Confirmed histopathologic diagnosis by National Cancer Institute (NCI) Laboratory of Pathology
* If tissue diagnosis is not feasible for any reason, such as undue risk to the patient to acquire tissue diagnosis, the following will be accepted as confirmed Acquired immunodeficiency syndrome-related primary central nervous system lymphoma (AR-PCNSL) diagnosis:
* Positive brain fluro-2-deoxy-d-glucose positron emission tomography (FDG-PET) and
* Epstein Barr Virus (EBV) detected in the cerebrospinal fluid (CSF) using polymerase chain reaction (PCR)
* Age 18 years or greater
* Eastern Cooperative Oncology Group (ECOG) performance less than or equal to 0-4
* Ability to understand and willing to provide informed consent
* If patient unable to understand informed consent, a previously designated durable power of attorney for healthcare or an individual with legal authority may substitute in this capacity
* Assignment of a durable power of attorney for healthcare if not already done

EXCLUSION CRITERIA:

* Prior therapy for central nervous system (CNS) lymphoma
* Steroids not an exclusion
* Evidence of lymphoma outside of the central nervous system
* Ocular involvement will not exclude
* Multidrug resistant HIV not amenable to long-term suppression based on either or both:
* Clinical history of poor adherence to multiple antiretroviral drugs deemed sufficient to render effective HIV control unattainable;
* HIV mutational analysis (genotyping and/or phenotyping) that reveals high-level resistance to more than 1 class of anti-HIV drugs such that a combination regimen comprised of agents from at least two drug classes can not be devised to suppress HIV long-term.
* Refusal to adhere to highly active antiretroviral therapy (HAART)
* Concurrent malignancy other than Kaposi sarcoma, resectable squamous cell or basal cell skin cancer, or T1 anal cancer amenable to surgical resection.
* Heart failure, Class IV by New York Heart Association criteria
* Chronic Liver Disease, Child-Pugh class B or C

Pregnancy

* Refusal to practice contraception during chemotherapy.
* Any condition or set of circumstances that the Principal Investigator or Protocol Chair interprets as creating undue risk to the patient by participating on this study or would make the patient unlikely to comply with the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09-14 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine AM. AIDS-related malignancies: the emerging epidemic. J Natl Cancer Inst. 1993 Sep 1;85(17):1382-97. doi: 10.1093/jnci/85.17.1382. PMID 8350362
- [Background] Goplen AK, Dunlop O, Liestol K, Lingjaerde OC, Bruun JN, Maehlen J. The impact of primary central nervous system lymphoma in AIDS patients: a population-based autopsy study from Oslo. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Apr 1;14(4):351-4. doi: 10.1097/00042560-199704010-00007. PMID 9111477
- [Background] von Gunten CF, Von Roenn JH. Clinical aspects of human immunodeficiency virus-related lymphoma. Curr Opin Oncol. 1992 Oct;4(5):894-9. doi: 10.1097/00001622-199210000-00012. PMID 1457504
- [Derived] Kranick SM, Goncalves PH, Stetler-Stevenson M, Aleman K, Polizzotto MN, Little RF, Yarchoan R, Uldrick TS. Paradoxical central nervous system immune reconstitution syndrome in acquired immunodeficiency syndrome-related primary central nervous system lymphoma. Haematologica. 2015 Jan;100(1):e21-4. doi: 10.3324/haematol.2014.114736. Epub 2014 Oct 10. No abstract available. PMID 25304612
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0051.html

RESULTS

PARTICIPANT FLOW:
Period: Induction Treatment
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Started | 12
Completed | 9
Not Completed | 3
Not completed — Died before completing. | 2
Not completed — Started induction w/MTX, RIX, & Temozol | 1
Period: Consolidation Treatment
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.74 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Median Baseline Mini Mental State Exam (MMSE) Score [Median (Full Range); unit: score on a scale] — The MMSE is scored out of a maximum of 30 points. A score of >25 is considered normal, with scores <25 indicating different levels of cognitive impairment: mild (21-24) moderate (10-20), and severe (0-10).
  score on a scale | 22 [5 to 29]
Median Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status [Median (Full Range); unit: scores on a scale] — ECOG Scale: 0 is fully active and able to carry on activities of daily living without restriction; 1 is restricted in physically strenuous activity but ambulatory, can perform light housework; 2 is ambulatory and able to perform self care but unable to carry out work activities; 3 is capable of limited self care and confined to bed or chair more than 50% of waking hours; 4 is completely disabled, unable to perform selfcare, and confined to bed or chair; and 5 is dead.
  scores on a scale | 2 [1 to 3]
Baseline Cluster of Differentiation (CD4) T Cell Count at PCNSL Diagnosis [Median (Full Range); unit: cells/µL] — Primary central nervous system lymphoma (PCNSL). PCNSL was biopsy confirmed or made by fludeoxyglucose positron emission tomography/cerebral spinal fluid Epstein Barr-Virus (EBV) viral load criteria.
  cells/µL | 16 [0 to 409]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive at 2 Years Without Recurrent Brain Lymphoma or Severe Neurocognitive Defects
Description: Recurrent lymphoma as defined by the International Primary Central Nervous System (CNS) Lymphoma Collaborative Group for response assessment of aggressive Non-Hodgkin's Lymphoma (NHL) using fluorodeoxyglucose F 18 (18FDG-PET). Severe cognitive problems are defined as the inability to carry out normal activities with minimal difficulty and not requiring nursing care or hospitalization because of neurological impairment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 12
Participants | 8

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 142 months and 11 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 12
Participants | 11

3. Secondary Outcome: Number of Participants With Response to Treatment After Rituximab, High-Dose Methotrexate (R-HD-MTX) Induction
Description: Response was assessed by the International Workshop Criteria for Non-Hodgkin's Lymphoma. Complete Response is disappearance of all enhancing lesions on magnetic resonance imaging of the brain. Partial Response is a reduction of enhancing tumor volume by more than 50% for at least 4 weeks. Progressive Disease is an increase of tumor volume of more than 25% or occurrence of new lesions.
Time Frame: At the end of 6 cycles or 12 weeks of treatment
Population: Two participants were not evaluable. One participant received one cycle of therapy and one was not evaluable due to treatment failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 10
Participants
  Complete Response | 5
  Partial Response | 4
  Progressive Disease | 1

4. Secondary Outcome: Estimated Percentage of Participants Overall Survival
Description: Participants that are estimated to be alive or last known to be alive after Rituximab, High-Dose Methotrexate and Leucovorin treatment.
Time Frame: Time from treatment start date until date of death or date last known alive, approximately 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 12
percentage of participants | 66 [32 to 86]

5. Secondary Outcome: Median Mini Mental Status Exam (MMSE) Score in Surviving Participants After Rituximab, High-Dose Methotrexate & Leucovorin ( R-HD-MTX) Treatment
Description: The MMSE is scored out of a maximum of 30 points. A score of >25 is considered normal, with scores <25 indicating different levels of cognitive impairment: mild (21-24) moderate (10-20), and severe (0-10).
Time Frame: up to 2.5 years
Population: as for outcome 3
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 10
Scores on a scale | 28 [27 to 30]

6. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) T Cell Count at up to 2.5 Years
Description: An increase in CD4 cells is determined by the number of CD4+ T lymphocytes /µL of peripheral blood.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 3
Measure: Median (Full Range); unit: cells/µL
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
Number analyzed (Participants) | 10
cells/µL | 35 [-54 to 369]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 142 months and 11 days.
Arm/Group | Rituximab, High-Dose Methotrexate & Leucovorin Treatment
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, High-Dose Methotrexate & Leucovorin Treatment (N=12)
Death not associated with CTCAE term::Death NOS (General disorders) | 1 (1)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 1 (1)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, Patient intubated) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, Pulmonary embolism) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab, High-Dose Methotrexate & Leucovorin Treatment (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 9 (58)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 11 (64)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 10 (72)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (39)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 2 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (12)
Blurred vision (Eye disorders) | 1 (2)
CD4 count (Blood and lymphatic system disorders) | 5 (19)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 2 (4)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (8)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (5)
Cognitive disturbance (Nervous system disorders) | 3 (6)
Confusion (Nervous system disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Constitutional Symptoms - Other (Specify, Concentration) (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 4 (7)
Decreased gait (Musculoskeletal and connective tissue disorders) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 2 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (10)
Fibrinogen (Blood and lymphatic system disorders) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal - Other (Specify, (+) stool crytosporidium) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (46)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 10 (79)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (Specify, HSV) (Infections and infestations) | 5 (9)
Infection - Other (Specify, Pneumonia) (Infections and infestations) | 1 (1)
Infection - Other (Specify, Pruritic warts) (Infections and infestations) | 1 (1)
Infection - Other (Specify, Staph infection) (Infections and infestations) | 1 (2)
Infection - Other (Specify, Stool Novovirus positive) (Infections and infestations) | 1 (1)
Infection - Other (Specify, Stool rotavirus) (Infections and infestations) | 1 (1)
Infection - Other (Specify, Urine culture positive) (Infections and infestations) | 1 (1)
Infection - Other (Specify, ) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 2 (3)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 11 (108)
Lymphopenia (Blood and lymphatic system disorders) | 8 (69)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9 (40)
Memory impairment (Nervous system disorders) | 4 (7)
Mood alteration::Agitation (Nervous system disorders) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1)
Mood alteration::Depression (Nervous system disorders) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Specify, Intermittent myoclonic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 1 (3)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10 (89)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1)
PCP Infection (Infections and infestations) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (2)
Pain - Other (Specify, BLE pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (Specify, Ear pain) (Ear and labyrinth disorders) | 1 (1)
Pain - Other (Specify, Left eye discomfort) (Eye disorders) | 1 (1)
Pain - Other (Specify, Thigh pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (Specify, Testicular pain) (Reproductive system and breast disorders) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 2 (4)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Oral-gums (Gastrointestinal disorders) | 1 (1)
Pain::Pain NOS (General disorders) | 1 (1)
Pain::Rectum (Gastrointestinal disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (15)
Platelets (Blood and lymphatic system disorders) | 9 (29)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 7 (14)
Proteinuria (Metabolism and nutrition disorders) | 3 (10)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Sleepy Somnolence (Nervous system disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 5 (15)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (12)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 (2)
Supraventricular and nodal arrhythmia::Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (2)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (2)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Ventricular arrhythmia::Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (General disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT00267865/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT00267865/ICF_001.pdf